CLINICAL TRIAL: NCT03492294
Title: The Role of Music Stimulation in Disorders of Consciousness State: an fMRI Study
Status: Completed | Type: Observational
Sponsor: Hangzhou Normal University (Other)
Responsible Party: Principal Investigator, Jing Wang, Dr, Hangzhou Normal University
Other Study IDs: 2008W1224
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Vegetative State; Minimally Conscious State
Keywords: disorders of consciousness; music stimulation; functional magnetic resonance imaging
MeSH Terms: conditions — Persistent Vegetative State; Consciousness Disorders | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with disorders of consciousness: patients with disorders of consciousness from several brain injury have been clinically classified into coma, unresponsive wakefulness syndrome and minimally conscious state. These patients were scaned by functional magnetic resonance imaging.
  Interventions: Diagnostic Test: functional magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: functional magnetic resonance imaging — Patients with disorders of consciousness were assessed by functional magnetic resonance imaging while they were exposed under the condition of music.
  Other Names: Coma Recovery Scale-Revised

SUMMARY:
The aim of the present study was to evaluated the neural effect of music on the cerebral activation in unresponsive wakefulness syndrome (UWS) and minimally conscious state (MCS) by using functional magnetic resonance imaging (fMRI).

DETAILED DESCRIPTION:
Background: Sensory stimulations were used widely to evaluate the preserved cerebral functions for these patients with disorders of consciousness. Among these, the most alerting or common stimuli are probably familiar voice and music.

Objective: The aim of the present study was to evaluated the neural effect of music on the cerebral activation in unresponsive wakefulness syndrome (UWS) and minimally conscious state (MCS) by using functional magnetic resonance imaging (fMRI).

Methods: Eleven severely brain-damaged patients (6 UWS and 5 MCS) were assessed by functional magnetic resonance imaging while they were exposed under the condition of their personal music. To examine the prognostic value of these patients, longitudinal behavioral assessments were repeatedly conducted by means of the CRS-R after fMRI acquisition.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years old;
* no administration of neuromuscular blockers or sedation within the 24 hours of enrolment;
* brain damage with eye opening (indicating wakefulness and rest cycles)

Exclusion Criteria:

* Coma;
* neurodegenerative disease;
* psychiatric or neurologic illness;
* with intracranial metal or other body metal.

Ages: 21 Years to 61 Years | Sex: All
Age Groups: Adult
Study Population: patients with disorders of consciousness
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Coma Recovery Scale-Revised | one to two years
  examine the prognostic value of these patients, longitudinal behavioral assessments were repeatedly conducted by means of the CRS-R after fMRI acquisition

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Di, Pro, Study Chair — International Vegetative State and Consciousness Science Institute, Hangzhou Normal University
Locations (1):
- International Vegetative State and Consciousness Science Institute, Hangzhou Normal University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Owen AM, Coleman MR. Detecting awareness in the vegetative state. Ann N Y Acad Sci. 2008;1129:130-8. doi: 10.1196/annals.1417.018. PMID 18591475